CLINICAL TRIAL: NCT00315900
Title: Depakote ER vs. Seroquel for Agitated Behaviors in Nursing Home Care Unit Patients With Dementia
Brief Title: Depakote Extended Release (ER) Versus Seroquel for Agitated Behaviors in Nursing Home Care Unit Patients With Dementia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Investigator closed study and left VAMC.
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Lori Davis, MD, Associate Chief of Staff for Research, Tuscaloosa Research & Education Advancement Corporation
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TREAC00081; 06-13 Station number (Other: Tuscaloosa VA IRB)
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Agitation; Dementia
Keywords: Seroquel; Depakote ER; Nursing Home; Quetiapine; Divalproex ER; Agitation
MeSH Terms: conditions — Psychomotor Agitation; Dementia | interventions — Valproic Acid; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Depakote ER (Experimental): Depakote ER
  Interventions: Drug: Depakote ER
- Seroquel (Active Comparator): Seroquel
  Interventions: Drug: Seroquel

INTERVENTIONS:
Drug: Depakote ER — depakote ER
  Other Names: Divalproex
  Arms: Depakote ER
Drug: Seroquel — seroquel
  Other Names: quetiapine
  Arms: Seroquel

SUMMARY:
The primary objective of the study is to assess the relative efficacy of Depakote ER and Seroquel for agitated behaviors among veterans with a dementia diagnosis residing in a Department of Veterans Affairs (VA) nursing home care unit (NHCU). The secondary objective of the study is to assess the relative tolerability of Depakote ER and Seroquel in this population. The primary hypothesis is that agitated dementia patients will demonstrate a significantly greater reduction in Cohen-Mansfield Agitation Inventory (CMAI) scores while treated with Depakote ER compared to treatment with Seroquel.

DETAILED DESCRIPTION:
This study is a prospective, single-center, randomized, double-blind, double-dummy, crossover trial of Depakote ER vs. Seroquel for agitated behaviors among veterans with dementia. After consent is obtained and after a washout period of one week or five half-lives after taper (if necessary), 20 eligible patients will be randomized to received one of two treatments. The first is DEPAKOTE ER, initiated at 250 mg daily. The other treatment will be Seroquel, starting at 25 mg BID. Both treatments will be co-administered with a placebo that matches the other drug (to preserve blinding). Using serial examinations and blinded laboratory reporting, doses will be adjusted to clinical response or to achieve a serum valproate level of at least 50 mcg/mL. After a treatment period of six weeks, patients will be crossed over to the other treatment without washout (doses will be adjusted concurrently) for a second six-week treatment period. The Cohen-Mansfield Agitation Inventory (CMAI) will be the primary outcome measure. Secondary measures include the Behavior Pathology in Alzheimer's Disease Rating Scale (BEHAVE-AD); Clinical Global Impression Scale - Severity; Clinical Global Impression Scale - Improvement; Barnes Akathisia Scale (BAS); and the Abnormal Involuntary Movements Scale (AIMS). Outcome measures will be performed at the end of each six-week treatment period to avoid carryover effects.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* Males or females
* Aged 55 or older
* With a diagnosis of dementia (either Alzheimer's disease, vascular dementia, or mixed Alzheimer's and vascular dementia)
* Residing in a Tuscaloosa VA Medical Center (TVAMC) NHCU bed
* Admitted to a NHCU bed at Tuscaloosa VA Medical Center
* Score of > 5 on the Functional Assessment Staging (FAST) scale
* Score of < 23 on the Mini-Mental State Examination
* Score of > 1 on the Behavior Pathology in Alzheimer's Disease Rating Scale (BEHAVE-AD) global rating
* Total BEHAVE-AD score of > 8
* Agitation present (by history or chart review) for at least two weeks (to minimize chance of enrolling for agitation due to delirium).

Exclusion Criteria:

* Diagnosis of dementia caused by a condition other than either Alzheimer's disease, vascular dementia, or mixed Alzheimer's and vascular dementia
* History of schizophrenia, bipolar disorder, or schizoaffective disorder
* Untreated depressive or anxiety disorder
* Untreated pain evident on physical examination
* Known allergy or hypersensitivity to either study drug
* History of epilepsy or seizures
* Diagnosis of liver disease or significant abnormalities on liver function tests
* Thrombocytopenia
* Diagnosis or past history of pancreatitis
* Past history of neuroleptic malignant syndrome
* Co-morbid condition that would render tapering off of current antipsychotics or anticonvulsants unsafe
* History of agitation unresponsive to an adequate previous trial of either valproate or quetiapine
* The patient has no identifiable guardian, decision-making proxy, or next of kin to approach for consent to participate.
* The patient's guardian, decision-making proxy, or next of kin withholds, or does not grant, consent to participate
* Patient judged to be too ill to participate

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2007-12-01 (Actual); Study Completion 2008-02-28 (Actual)

PRIMARY OUTCOMES:
Cohen-Mansfield Agitation Inventory (CMAI) | 12 week
  Cohen-Mansfield Agitation Inventory (CMAI) is a 29-item scale to systematically assess agitation (higher is more severe).

SECONDARY OUTCOMES:
Behavioral Pathology in Alzheimer's Disease Rating Scale (BEHAVE-AD) | 12 weeks
  A psychiatric rating scale to evaluate behavioral disturbances in dementia patients. assesses 25 potentially remediable behavioral symptoms on a 4-rating-point severity scale (higher score is more severe).

CONTACTS AND LOCATIONS:
Overall Officials: John L Shuster, MD, Principal Investigator — Tuscaloosa Veterans Affairs Medical Center
Locations (1):
- Tuscaloosa VA Medical Center, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shuster JL Jr. Palliative care for advanced dementia. Clin Geriatr Med. 2000 May;16(2):373-86. doi: 10.1016/s0749-0690(05)70062-8. PMID 10783434